CLINICAL TRIAL: NCT04497454
Title: Mechanical Ventilation Strategy for Coronavirus Disease 2019 (COVID-19) - COVEN Study
Brief Title: Mechanical Ventilation Strategy for Coronavirus Disease 2019 (COVID-19)
Acronym: COVEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 30938720800000068
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Distress Syndrome; Mechanical Ventilation; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center, open-label, superiority, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARDSNet (Active Comparator): ARDSNet protocol (low PEEP-FiO2 table). Ventilatory mode: volume-controlled ventilation Tidal volume (VT) will be adjusted to 4-6 mL/Kg of PBW and Plateau pressure < 30 cmH2O for the at least the first 12 hours after inclusion in the protocol pH should be maintained between 7.35-7.45 Oxygenation (SpO2) target ranges 90-95% Maximum respiratory rate = 35 breaths/min PEEP and FIO2 adjusted according to the low PEEP-FiO2 Table.
  Interventions: Other: ARDSNet
- EIT-Group (Experimental): The goal is to maintain driving pressure (DP) < 16 cmH2O. Ventilatory mode: pressure-controlled ventilation After a recruitment a maneuver, PEEP will be chosen according to a PEEP titration maneuver monitored with electrical impedance tomography Plateau pressure may exceed 30 cmH2O and VT may exceed 6 mL/Kg if DP < 16 cmH2O pH should be maintained between 7.15-7.40 Oxygenation (SpO2) target ranges 90 -95% Maximum respiratory rate = 50 bpm
  Interventions: Other: EIT-Group

INTERVENTIONS:
Other: EIT-Group — A mechanical ventilation strategy with the main goal to maintain DP < 16 cmH2O
  Arms: EIT-Group
Other: ARDSNet — Low PEEP-FiO2 table ARDS Network ventilation protocol
  Arms: ARDSNet

SUMMARY:
This is a prospective, randomized, single-center, open-label controlled trial, designed to compare the efficacy of two ventilation strategies (Low Tidal Volume and positive end-expiratory pressure (PEEP) based on the Acute Respiratory Distress Syndrome (ARDS) Network low PEEP-fraction of inspired oxygen inspired oxygen fraction (FIO2) Table versus Low Driving Pressure and PEEP guided by Electrical Impedance Tomography (EIT) in reducing daily lung injury score in patients with acute respiratory distress syndrome caused by COVID-19. The two strategies incorporate different prioritizations of clinical variables. The PEEP-FIO2 table strategy aims to reduce lung overdistension, even if it requires tolerating worse gas exchange. EIT-guided strategy prioritizes mechanical stress protection, avoiding alveolar overdistension and collapse.

DETAILED DESCRIPTION:
Mechanical ventilatory strategy of the ARDS Network low PEEP-FiO2 table will be followed in the control arm. This strategy consists of at least 12 hours of controlled mechanical ventilation following prespecified PEEP and FiO2 combinations chosen dynamically targeting oxygenation. Tidal volume is set at 4-6 mL/Kg of predicted body weight (PBW) and plateau pressure is kept below 30 centimeters of water (cmH2O). Respiratory rate can be as high as 35 breaths per minute titrated to a potential of hydrogen (pH) 7.30-7.45. As oxygenation improves, patients are transitioned to assisted ventilation and then to pressure support ventilation until they are ready to be liberated from the ventilator. During this phase, no attempt is made to control plateau pressures or tidal volumes. In the intervention arm, minimizing tidal lung strain by keeping driving pressure below 16 cmH2O throughout the mechanical ventilation period will be targeted. The controlled phase will last at least 48 hours. PEEP will be selected according to a PEEP titration maneuver with EIT at the start of the intervention. This PEEP level will be kept until extubation. Respiratory rate can be as high as 50 breaths per minute targeting a pH of 7.15-7.45.

ELIGIBILITY:
Inclusion Criteria:

Patients under mechanical ventilation with ARDS (Berlin definition) caused by SARS-COV2 infection:

* ARDS diagnosis in less than 24 hours
* Respiratory System Compliance of 0.6 mL/cmH2O/Kg of PBW

Exclusion Criteria:

* Age < 18 years
* Active bronchopleural fistula
* History of chronic and disabling respirator disease, requiring home oxygen treatment
* Chronic pulmonary arterial hypertension (pulmonary artery systolic pressure > 40 mmHg)
* Huge intrathoracic tumoral mass
* Electrical impedance tomography monitoring contraindications (as thoracic wounds or burns, electronic implantable devices)
* Hemodynamic instability (systolic pressure < 80 mmHg or mean arterial pressure < 60 mmHg, despite vasopressor drugs; and/or heart rate < 55bpm) - this patient may be included after recovered from hemodynamic instability
* Not drained pneumothorax or subcutaneous emphysema or bronchopleural fistula
* Patients at risk of intracranial hypertension development or post Cardiopulmonary resuscitation (first 72 hours)
* Pregnancy
* Impossibility of monitoring with EIT
* Not committed to full support or life expectation < 24 hours
* Legal responsible or clinical team refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Average daily Modified Lung injury score until day 28 | daily
  This score originally ranges from 0 to 4 points based on the average of 4 parameters (PaO2/FiO2, chest X-Ray, PEEP level, and Respiratory compliance). In the modified version, if the patient dies, he or she automatically receives a score of 5 irrespective of the other four parameters. If the patient is extubated, the score is automatically zero. We also substituted FiO2 for PEEP guaranteeing equivalence of the score when either the low or high PEEP-FiO2 table is applied.

SECONDARY OUTCOMES:
High oxygen dependence free days until day 28 | 28 days
  Number of days with less than or equal to 1 Liter/min of oxygen supplementation until day 28
Mechanical ventilation free days until day 28 | 28 days
  Number of days free of mechanical ventilation assistance after protocol inclusion and before day 28
Incidence of shock or barotrauma | 28 days
  Occurrence of shock (persistent hypotension despite rescue measures) and incidence of barotrauma
Incidence of acute renal failure requiring renal replacement therapy | 28 days
  Occurrence of acute renal failure that justifies renal replacement therapy
28-day mortality | 28 days
  Percentage of patients who died in each arm up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo LV Costa, PhD, Principal Investigator — Hospital das Clinicas from University of São Paulo
Locations (1):
- USP Instituto do Coração, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa ELV, Alcala GC, Tucci MR, Goligher E, Morais CC, Dianti J, Nakamura MAP, Oliveira LB, Pereira SM, Toufen C Jr, Barbas CSV, Carvalho CRR, Amato MBP. Impact of extended lung protection during mechanical ventilation on lung recovery in patients with COVID-19 ARDS: a phase II randomized controlled trial. Ann Intensive Care. 2024 Jun 8;14(1):85. doi: 10.1186/s13613-024-01297-z. PMID 38849605
- [Derived] Hohmann F, Wedekind L, Grundeis F, Dickel S, Frank J, Golinski M, Griesel M, Grimm C, Herchenhahn C, Kramer A, Metzendorf MI, Moerer O, Olbrich N, Thieme V, Vieler A, Fichtner F, Burns J, Laudi S. Early spontaneous breathing for acute respiratory distress syndrome in individuals with COVID-19. Cochrane Database Syst Rev. 2022 Jun 29;6(6):CD015077. doi: 10.1002/14651858.CD015077. PMID 35767435